CLINICAL TRIAL: NCT05245617
Title: A Single Center Post-market Clinical Follow up (PMCF) Observational Study Evaluating the Clinical Performance and the Safety Profile of the JuniOrtho™ Plating System™ (JPS) for the Treatment of Congenital Deformities and Fractures in Lower Limb of Pediatric and Adult Patients
Brief Title: Observational Study on JuniOrtho Plating System for Deformities and Fractures Treatment in Lower Limb
Acronym: JPS
Status: Completed | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2102
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Deformity; Defect, Congenital; Trauma
Keywords: Femur; Tibia; Congenital; deformity; Plate; Fracture
MeSH Terms: conditions — Congenital Abnormalities; Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JPS treated patients: This grup will include all patients with regular indication for JPS: system is intended in pediatric (excluding newborns) and small stature adult patients. Pediatric patients include infants (greater than 1 month to 1 years of age), children (greater than 1 to 12 years of age), adolescents (greater than 12 to 18 years of age) and appropriate adults (where according to investigator assessment, the JPS plates fit the treated bone anatomy).
  Interventions: Device: JuniOrtho™ Plating System™

INTERVENTIONS:
Device: JuniOrtho™ Plating System™ — The patient underwent surgery for the application of JPS for treatment of deformity or traumatic fracture.
  Other Names: JPS

SUMMARY:
Orthofix Srl put the JPS on the European market (2019) by the mean of a pre-market clinical evaluation made under the Medical Device Directive (MDD) requirements that were based on the analysis of the scientific literature of equivalent devices.

This study has been planned as part of the Orthofix Srl post-market active surveillance plan for the collection of data on both the clinical performance and the safety profile of the JPS in a representative population of Patients and users.

The rationale of the proposed study is to update and support the pre-market clinical evaluation of the JPS with real-word-evidence clinical data, in order to confirm the benefit/risk ratio of this medical device and to keep the CE mark under Medical Device Regulation (MDR) requirements.

DETAILED DESCRIPTION:
One selected site that is experienced in the treatment of pediatric and adult patients with bone deformities and fractures, where the usage of JPS is already part of the normal clinical practice, will participate in this study. Investigator will provide data for a maximum of 40 JPS implant cases satisfying inclusion and exclusion criteria (predicted drop out rate is 10%) that will contribute for at least 30 cases treated by JPS (note that some patients may contribute for more than one JPS case, according to how many JPS implants were received).

For retrospective study cohort, who has previously had JPS implanted and follow-up assessment and JPS removal is done, the investigators shall purely collect clinical data from the medical record of the subjects, concerning the screening criteria, the surgery (MD application) and 4 following events: hospital discharge, first post-application control, bone consolidation assessment and device removal. Data from patients' observation are collected according to the site standard-of-care.

Patients, who are prospectively enrolled in the study and have undergone JPS implantation, will have follow-up assessments, as described on Table 10.2, or until patient withdrawal.

The patient data will be systematically collected by the investigator in eCRF. As per CIP, the subjects will not undergo additional visit nor non-invasive, invasive or burdensome procedures additional to those performed under the normal clinical practice.

ELIGIBILITY:
Inclusion Criteria: a patient will be eligible for inclusion in the study if:

* had a regular indication for surgical intervention with JPS according to the manufacturer's IFU;
* underwent a surgery for bone deformity correction or trauma reconstruction of the lower extremities performed by JPS;
* the clinical data registered in her/him patient chart are sufficient to assess the safety and efficacy endpoint of the study;
* patient (or his/her legally acceptable representative) is capable of understanding the content of the Informed Consent Form (ICF) [applicable for the prospective group of patients]
* patient is willing and able to participate in the prospective data collection and comply with the protocol requirements;

Note: for the retrospective group of patients to whom all interventions and control visits were already done, a waiver of consent for retrospective data collection to be requested.

Exclusion Criteria: a Patient will be excluded from participation in the study if he/she:

* had/has a medical condition that is a contraindication according to the manufacturer's instruction for use leaflet;
* had/has a concomitant not permitted device which cannot be safely removed;
* patient for whom there are other concurrent medical or other conditions that in opinion of the participating investigator may prevent participation or otherwise render patient ineligible for the study.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted only on patients with a regular indication for JPS JuniOrtho Plating System as per IFU: the system is intended in pediatric (excluding newborns) and small stature adult patients. Pediatric patients include infants (greater than 1 month to 1 years of age), children (greater than 1 to 12 years of age), adolescents (greater than 12 to 18 years of age) and appropriate adults (where according to investigator assessment, the JPS plates fit the treated bone anatomy).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Leidinger, MD, Principal Investigator — Orthopädische Klinik Volmarstein
Locations (1):
- Orthopädische Klinik Volmarstein, Wetter, Ruhr, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joeris A, Audige L, Ziebarth K, Slongo T. The Locking Compression Paediatric Hip Plate: technical guide and critical analysis. Int Orthop. 2012 Nov;36(11):2299-306. doi: 10.1007/s00264-012-1643-1. Epub 2012 Aug 26. PMID 22923267
- [Background] Sidler-Maier CC, Reidy K, Huber H, Dierauer S, Ramseier LE. LCP 140 degrees Pediatric Hip Plate for fixation of proximal femoral valgisation osteotomy. J Child Orthop. 2014 Feb;8(1):29-35. doi: 10.1007/s11832-014-0550-y. Epub 2014 Jan 28. PMID 24488843
- [Background] Masquijo JJ. Percutaneous plating of distal tibial fractures in children and adolescents. J Pediatr Orthop B. 2014 May;23(3):207-11. doi: 10.1097/BPB.0000000000000036. PMID 24500423
- [Background] Xu Y, Bian J, Shen K, Xue B. Titanium elastic nailing versus locking compression plating in school-aged pediatric subtrochanteric femur fractures. Medicine (Baltimore). 2018 Jul;97(29):e11568. doi: 10.1097/MD.0000000000011568. PMID 30024559
- [Background] Islam SU, Henry A, Khan T, Davis N, Zenios M. The outcome of paediatric LCP hip plate use in children with and without neuromuscular disease. Musculoskelet Surg. 2014 Dec;98(3):233-9. doi: 10.1007/s12306-013-0308-6. Epub 2013 Dec 3. PMID 24297691
- [Background] Zheng P, Yao Q, Xu P, Wang L. Application of computer-aided design and 3D-printed navigation template in Locking Compression Pediatric Hip PlateTauMu placement for pediatric hip disease. Int J Comput Assist Radiol Surg. 2017 May;12(5):865-871. doi: 10.1007/s11548-017-1535-3. Epub 2017 Feb 11. PMID 28190127

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: implants (i.e. procedures)
Period: Overall Study
Arm/Group | JPS Treated Patients
Started | 30; 46 implants (i.e. procedures)
Completed | 29; 44 implants (i.e. procedures)
Not Completed | 1; 2 implants (i.e. procedures)
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | JPS Treated Patients
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at surgery | 19.9 (6.3)
  Age at ICF signature | 21.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Subjects With at Least One Serious/Not Serious Adverse Event Certainly Related or Possibly Related to JPS (ADEs)
Description: Percentage of subjects who experience at least one adverse event (serious or non-serious) that the investigator judges as certainly or possibly related to the JPS system (ADEs). This outcome is used to assess the safety profile of the JPS system.
Time Frame: Up to 18 months from surgery (at device removal)
Measure: Number (95.2% Confidence Interval); unit: percentage of subjects
Arm/Group | JPS Treated Patients
Number analyzed (Participants) | 30
percentage of subjects | 3.3 [0.1 to 17.4]

2. Primary Outcome: Percentage (%) of Subjects With at Least One Medica Device Deficiencies (MDDs)
Description: Percentage of subjects who experienced at least one medical device deficiency (MDD) i.e., any inadequacy, malfunction, or nonconformance of the investigational device or its accessories, during the defined observation window. This outcome is used to asses the safety profile of the JPS system.
Time Frame: Up to 18 months from surgery (at device removal)
Measure: Number (95.2% Confidence Interval); unit: percentage of subjects
Arm/Group | JPS Treated Patients
Number analyzed (Participants) | 30
percentage of subjects | 70.0 [50.4 to 85.4]

3. Secondary Outcome: Percentage (%) of Subjects That Reached a Satisfactory Bone Consolidation According to Investigator's Opinion
Description: Percentage of subjects who achieved satisfactory bone consolidation, as judged by the investigator per protocol-defined criteria, up to the specified assessment time point. This outcome is used to asses the clinical performance of the JPS system.
Time Frame: Up to 18 months from surgery (at device removal)
Measure: Number (95.2% Confidence Interval); unit: percentage of subjects
Arm/Group | JPS Treated Patients
Number analyzed (Participants) | 30
percentage of subjects | 96.7 [82.6 to 99.9]

4. Secondary Outcome: Percentage (%) of Subjects That Maintained Bone Correction Alignment According to Investigator's Opinion
Description: Percentage of subjects who maintained bone correction alignment, as assessed by the investigator per protocol-defined criteria, up tp the specified follow-up time point. Note: This outcome is calculated only for the subgroup "JPS-Treated Patients for Deformity Correction.", that is the only patients that present a correction alignment. This outcome is used to asses the clinical performance of the JPS system.
Time Frame: Up to 18 months from surgery (at device removal)
Measure: Number (95.2% Confidence Interval); unit: percentage of subjects
Groups:
- JPS-Treated Patients for Deformity Correction: This subgroup consists of patients enrolled in the study who were treated with the JPS medical device specifically for deformity correction. Patients treated with JPS for fractures or other indications were excluded, as they did not undergo a corrective alignment procedure.
Arm/Group | JPS-Treated Patients for Deformity Correction
Number analyzed (Participants) | 27
percentage of subjects | 96.3 [80.9 to 99.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from treatment through the last available follow-up for each patient, with a maximum follow-up duration of up to 18 months, in accordance with site standard practice.
Description: For the retrospective cohort, collect only AEs and MDDs already in medical files from application to device removal. For the prospective cohort, follow clinical practice, CA reporting, and manufacturer instructions before recording AEs/MDDs in the eCRF. In both cohorts, when reporting in eCRF, assess seriousness and device relation. From surgery to removal, record AEs in the patient eCRF as appropriate.
Arm/Group | JPS Treated Patients
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JPS Treated Patients (N=30)
Delayed union, nonunion, malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Events caused by anesthesia and surgery (Surgical and medical procedures) | 1 (1)
Loosening of the implant and loss of fixation (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JPS Treated Patients (N=30)
Events caused by anesthesia and surgery (Surgical and medical procedures) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor and investigator may publish or present study results, submit data to regulatory authorities, and register the study publicly. Co-authors may submit manuscripts/abstracts to the sponsor for review before publication. Sponsor's proposed changes must not affect scientific content. The sponsor's identity and contribution must be disclosed in all publications or presentations.

DOCUMENTS (2):
  • Study Protocol (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT05245617/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT05245617/SAP_001.pdf